CLINICAL TRIAL: NCT03925051
Title: A Randomized, Double-masked, Parallel-group Study, to Compare Pharmacokinetics, Safety and Immunogenicity of CMAB807 Injection Versus Prolia® in Healthy Chinese Male Subjects.
Brief Title: Phase 1 Study to Compare CMAB807 Injection to Prolia® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Biomabs Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB807-I-001
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: Randomized, Double-masked, Parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: subjects, investigator, sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMAB807 (Experimental): 60mg by subcutaneous injection once on the first day.
  Interventions: Drug: CMAB807
- Prolia® (Active Comparator): 60mg by subcutaneous injection once on the first day.
  Interventions: Drug: Prolia®

INTERVENTIONS:
Drug: Prolia® — mAb targeting RANKL. human monoclonal antibody targeting RANKL.
  Other Names: Denosumab Injection
  Arms: Prolia®
Drug: CMAB807 — human monoclonal antibody targeting RANKL.
  Other Names: Denosumab Injection
  Arms: CMAB807

SUMMARY:
CMAB807 is a human monoclonal antibody targeting the key bone resorption mediator RANKL. The drug is administered via subcutaneous injection once six months and is approved for various indications, including the treatment of postmenopausal women with osteoporosis at increased/high risk of fracture. This phase 1 clincical study investigates the pharmacokinetics, safety and immnogenicity of CMAB807,compared to prolia®, in healthy Chinese male subjects.

DETAILED DESCRIPTION:
This is a phase 1 single center, randomized, double-masked, parallel-group clinical trial. The primary objective is to assess the pharmacokinetics similarity of single and subcutaneous injection of CMAB807 injection or Prolia® in health volunteers. The secondary objectives are to assess the clinical safety and immnogenicity similarity of single and subcutaneous injection of CMAB807 or Prolia® in healty volunteers. Meanwhile, exploring the pharmacodynamic similarities of CMAB807 and Prolia®.

Subjects will receive a single 60mg of CMAB807 or Prolia® through subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntary sign the informed consent form,and be able to complete the study according to the protocol;
* 18 years ≤ age ≤65 years;
* Physical examination, vital signs, clinical laboratory examination and various examinations are normal or abnormal without clinical significance;
* Agree to take effective contraceptive measures throughout the study period (including not limited to: physical contraception, hormonal drugs of pregnancy, surgery, abstinence, etc.,) until at least 10 months after the last study is administered;
* Body weight ≥50 kg, 19kg/m2≤BMI≤26kg/m2;
* Serum calcium level between 2.15~2.55mmol/L（including the boundary value）;
* Normal or clinically acceptable electrocardiogram (12-lead ECG), QTcB<450msec.

Exclusion Criteria:

* Drink 14 units of alcohol per week within 3 months prior to administration, or take any alcohol substance within 48 hours before subcutaneous injection;
* Substance abuse within 5 years before subcutaneous injection;
* Smoke more than 5 cigarettes per day or the same amount of tobacco within 3 months before subcutaneous injection;
* Allergic constitution;
* Drink excessive amounts of tea, coffee or caffeinated beverages within 30 days before subcutaneous injection;
* Use any prescription, over-the-counter, vitamin or herbal medicine within 30 days before subcutaneous injection;
* Bone surgery was performed within 30 days before administration;
* History of osteomyelitis or osteonecrosis of the jaw;
* Inflammation or abnormalities in or around the site of administration;
* Needle or blood sickness;
* Dental disease or jaw disease requiring oral surgery, dental surgery; or plan to have dental surgery during the study;
* Received the study drug(including Xgeva and Prolia), or participated in a clinical trial within 3 months prior to administration；
* Received living viraL vaccine within 3 months prior to administration;
* Blood donation or blood loss >400ml within 3 months prior to administration;
* Hepatitis B surface antigen was positive, and/or hepatitis C antibody was positive;
* The HIV antibody test was not negative;
* Syphilitic test was positive;
* Drug was detected in the urine;
* Hyperparathyroidism, hypothyroidism, rheumatoid arthritis, Ankylosing Spondylitis, osteomalacia, Paget's disease, or fracture within 6 months;
* History of severe lumbar disc herniation;
* Insanity or legal problem are exist;
* Plan to engage in strenuous physical labor or exercise during the study;
* Other conditions that made it difficult to participate the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
AUC0-t | 0~126 day
  Area Under Curve(AUC)0-t
Cmax | 0~126 day
  Maximum Concentration

SECONDARY OUTCOMES:
Incidence of Adverse Event | 0~126 day
  measured by common terminology criteria for adverse events grading
Antidrug Antibody | 0~126 day
  Percentage of Subjects Positive for Antidrug Antibody
Serum type 1 C-telopeptide(CTX1) | 0~126 day
  explore the pharmacodynamic profile by detect the serum concentration of CTX1

CONTACTS AND LOCATIONS:
Overall Officials: xuening li, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Chen W, Yuan F, Guo Q, Zhang X, Wang C, Li X. Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of CMAB807, a New Denosumab Biosimilar, in Healthy Chinese Subjects. Front Pharmacol. 2022 Jan 24;13:821944. doi: 10.3389/fphar.2022.821944. eCollection 2022. PMID 35140619